CLINICAL TRIAL: NCT00984828
Title: A Randomized Study of 4 vs. 8 Cycles of Velcade-based Regimen With Autologous Stem Cell Transplantation in Newly-diagnosed Myeloma Patients
Brief Title: Randomized Study of Velcade-based Regimen With Autologous Stem Cell Transplantation in Newly-diagnosed Myeloma Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Very slow recruitment
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood and Marrow Transplantation Center, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMY3024
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; autologous stem cell transplantation; velcade
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vel 8 - ASCT (Experimental): 8 cycles of velcade with ASCT
  Interventions: Drug: velcade
- vel4 - ASCT (Active Comparator): 4 cycles of velcade with ASCT
  Interventions: Drug: velcade

INTERVENTIONS:
Drug: velcade — velcade 1.3mg/m2 D1, 4, 8 and 11
  Other Names: bortezomib

SUMMARY:
The is a randomized control study for newly-diagnosed myeloma patients 18-65 year old. All patients will receive 4 cycles of velcade and Dexamethasone as front-line therapy. Then patients will be randomized into standard group which will receive a single autologous hematopoietic stem cell transplantation with standard conditioning of melphalan 200mg/m2 and the study group which will receive single autologous hematopoietic stem cell transplantation with conditioning of melphalan 200mg/m2 + velcade followed by 3 more cycles of velcade alone as consolidation.

DETAILED DESCRIPTION:
The is a randomized control study for newly-diagnosed myeloma patients 18-65 year old. Newly-diagnosed myeloma patient enrolled will receive 4 cycles of velcade and Dexamethasone as front-line induction therapy. All patients finished the induction therapy will be randomized into standard group and the study group. All patients will mobilized by cyclophosphamide with G-CSF to collect a target of 2x106 CD34+/kg and then undergo autologous stem cell transplantation. For standard group, patients will receive single auto-SCT with standard conditioning of melphalan 200mg/m2. The patients in the study group will receive single auto-SCT with conditioning of melphalan 200mg/m2 added with 4 dose of velcade at 1.0mg/m2 during the transplantation procedure and then followed by 3 more cycles of velcade alone as consolidation.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between age 18-65 with newly diagnosed Multiple Myeloma for whom stem cell transplantation is considered appropriate
* Measurable serum and/or urinary paraprotein
* European Cooperative Oncology Group performance status 0-3
* Serum bilirubin < 1.5x the upper limit of normal (ULN) Serum alanine transaminase (ALT)/aspartate transaminase values < 2.5 x ULN
* Subjects (or their legally acceptable representatives) must signed an informed consent document indicating that they understanding the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Woman of child bearing potential
* Non-secretory MM
* Serum creatinine > 400 Micromol/l after initial resuscitation patients with previous Grade 2-4 peripheral neuropathy
* Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug)
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, uncontrolled angina, clinically significant pericardial disease, or III-IV heart failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-08; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 60 days and 2 years after the treatment

SECONDARY OUTCOMES:
Progression-free survival | 2 years
Overall survival | 2 years
Quality of life | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Xiang Shen, M.D., Principal Investigator — Rui Jin Hospital, Shanghai JiaoTong University School of Medicine
Locations (1):
- Rui Jin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No